CLINICAL TRIAL: NCT06535191
Title: Evaluating an Employment-related Social Skills Training Program for Transition-Age Youth With Autism (The ASSET Program): A Randomized Controlled Trial Study
Brief Title: The ASSET Program for Youth With ASD
Acronym: ASSET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: Illinois Institute of Technology (Other)
Responsible Party: Principal Investigator, Connie Sung, Professor, Michigan State University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000097
Record Dates: First submitted 2024-07-15; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Social Skills; Transition; Autism Spectrum Disorder; Confidence, Self
Keywords: Soft Skills; Work-related Social Skills; Autism Spectrum Disorder; School-to-work Transition; Vocational Rehabilitation; Employment
MeSH Terms: conditions — Social Skills; Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: The study uses a factorially designed randomized controlled trial [2 conditions (treatment vs. waitlist) x 3 intervals pre-, post-, 3-month follow-up].
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASSET Intervention (Experimental): Participants in the intervention group received Assistive Soft Skills and Employment Training (ASSET), a 10-week manualized soft skills intervention program to help students with ASD improve social and adaptive functioning, self-efficacy, work readiness, and anxiety.
  Interventions: Behavioral: Assistive Soft Skills and Employment Training (ASSET)
- Treatment As Usual (No Intervention): Participants in the treatment-as-usual is considered as control group and received typical education program.

INTERVENTIONS:
Behavioral: Assistive Soft Skills and Employment Training (ASSET) — ASSET program is a manualized, theory-driven, 10-week soft skills intervention for autistic individuals, who seek employment or who wish to maintain employment by improving work-related social skills. Throughout a 10-week curriculum offered in a school-based group setting, ASSET addresses the following competencies for workplace success: Communication, Networking, Enthusiasm and Attitude, Teamwork, Problem-Solving and Critical Thinking, Professionalism, Mental Health and Stress Management, and Awareness of Self and Others.
  Arms: ASSET Intervention

SUMMARY:
The purpose of this project is to evaluate the effectiveness of a work-related social skills training intervention for transition-age youth with Autism Spectrum Disorder (ASD; ages 14-22) that is designed to improve social skills, social self-efficacy, adaptive functioning, anxiety and work readiness. The Assistive Social Skills & Employment Training (ASSET) program is a weekly after-school program that runs for 10 weeks. In the first part of the study, youth with ASD, caregivers, special education teachers and employment specialists are invited to review and provide recommendations to improve the manual that has been developed for the ASSET program. The second part of the study is to evaluate the impact of the ASSET program on helping students with ASD improve their social skills, social self-efficacy, adaptive functioning, anxiety and work readiness using a randomized control trial. Improvements in these domains will be assessed immediately following the 10-week program and 3 months later. The intervention will occur at multiple sites in Michigan and Illinois, with a total of 96 students with autism. The ASSET program addresses the employment disparities faced by young adults with ASD by specifically targeting work-related social skills through the development of social skills and self-efficacy to foster successful school-to-work transition outcomes. The manualized ASSET program curriculum will eventually be made public and available for schools and service providers to use.

DETAILED DESCRIPTION:
Objective/Hypotheses: The objective of the randomized controlled trial (RCT) study is to evaluate the effectiveness of a manualized work-related social skills training intervention for transition-age youth (14-26 years old) with ASD designed to improve social skills and self-efficacy. The Assistive Social Skills and Employment Training (ASSET) program is a manualized 10-week program for 4-6 students with ASD that meets after school for 90 minutes on a weekly basis focusing on building work-related social skills for transition-age youth with ASD. It is hypothesized that students with ASD will show significantly greater improvements in social skills and social self-efficacy (primary outcomes) as well as adaptive functioning, anxiety and job readiness (secondary outcomes) compared to those in the waitlist control groups (a) at the end of the 10-week of the intervention and (b) at 3-month follow up.

Specific aims: First, the pilot-tested ASSET manual will be refined and finalized using community-based participatory action research (CBPR) approach gathering input from key stakeholder groups. Second, the effectiveness and sustainability of the ASSET program will be evaluated using a factorially designed randomized controlled trial [2 conditions (treatment vs. waitlist) x 3 intervals pre-, post-, 3-month follow-up].

Study Design: The first stage of this project incorporates stakeholder recommendations using a CBPR approach to refine the manual for the ASSET intervention. The second and third stages examine the efficacy of the ASSET program at immediate and follow-up using a randomized control trial design in two Midwestern states with randomization of student participants by condition for each of the two states, with a total of 4 treatment cycles over years 2 and 3 of the four-year study period, including 3-month follow-up after the completion of the 10-week program. Participants will include 96 students (age 14-22) from schools in Michigan and Illinois who will be randomly assigned to either the ASSET intervention or waitlist-control condition.

Clinical Impact: This project will fill an important gap for schools, transition providers, families and students, by testing an intervention designed to specifically improve the social functioning and self-efficacy of youth with ASD to improve work-related success. The findings will provide an empirically supported intervention manual to help students with ASD improve social and adaptive functioning, self-efficacy, work readiness, and anxiety.

ELIGIBILITY:
Inclusion Criteria:

1. aged between 14-22 years of age;
2. have a diagnosis of autism without intellectual disabilities (i.e., autistic disorders, Asperger's syndrome, PDD-NOS, Rett's syndrome, Childhood Disintegrative Disorder according to DSM-IV or Autism Spectrum Disorder according to DSM 5);
3. exhibit social problems as reported by self or caregiver.

Exclusion Criteria:

1. have a co-occurring intellectual disability;
2. have other neurological disorders or severe psychiatric disabilities.

Ages: 14 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 85 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-05-22 (Actual)

PRIMARY OUTCOMES:
Social Functioning | Pre-intervention, immediately post-intervention, 3-month post-intervention
  Social composite score of the Adaptive Behavior Assessment System: Third Edition (ABAS-3) was used to assess participants' changes in social functioning.
  Raw Scores: Each item within the Social Skills subdomains is rated on a 4-point Likert scale, ranging from 0 (Never) to 3 (Always). The ratings are summed to produce raw scores for each subdomain.
  Scaled Scores: Raw scores are converted to scaled scores for Social Skills subdomain. Scaled scores typically range from 1 to 19, with a mean of 10 and a standard deviation of 3.
  Composite Score: The scaled scores from the Social Skills subdomains are combined to form the Social Composite Score, with a mean of 100 and a standard deviation of 15, with a higher score indicating higher social functioning.
Social Responsiveness | Pre-intervention, immediately post-intervention, 3-month post-intervention
  Total score of the Social Responsiveness Scale: Second Edition (SRS-2) was used for measuring social responsiveness.
  Raw Scores: Each item is rated on a 4-point Likert scale, ranging from 0 (Never True) to 3 (Almost Always True). Raw scores are summed for each subscale and for the total scale. Subscales include: (1) Social Awareness; (2) Social Cognition; (3) Social Communication; (4) Social Motivation; and (5) Restricted Interests and Repetitive Behaviours.
  T-Scores: Raw scores are converted to T-scores to facilitate interpretation. T-scores have a mean of 50 and a standard deviation of 10, with a higher score indicating greater severity of social impairment.
Work Behaviors | Pre-intervention, immediately post-intervention, 3-month post-intervention
  Subscale scores of the Job Observation and Behavior Scale (JOBS) was used to assess participants' changes in work readiness and behaviors.
  Raw Scores: Each item is rated on a Likert scale. Individual item scores are summed to create raw scores for various subscales, which include (1) Work Quality, (2) Work Quantity, (3) Work Attitudes, (4) Social Skills, (5) Personal Presentation, and (6) Adaptability.
  Composite Scores: Raw scores from the subscales are combined to form composite scores (i.e., Quality of performance and Type of support), with a higher composite score indicating better performance, more positive work behaviors, less support/assistance needed.
Social Self-efficacy | Pre-intervention, immediately post-intervention, 3-month post-intervention
  Score of Perceived Social Self-Efficacy (PSSE) was used to assess participants' changes in perceived social self-efficacy. It is scored using a 5-point Likert scale, ranging from 1 (Not well at all) to 5 (Very well).
  The overall range of possible scores is 6 to 30, with a higher score indicating a higher level of social self-efficacy.
Empathic Self-efficacy | Pre-intervention, immediately post-intervention, 3-month post-intervention
  Score of Perceived Empathic Self-Efficacy (PESE) was used to assess participants' changes in perceived empathic self-efficacy. It is scored using a 5-point Likert scale, ranging from 1 (Not well at all) to 5 (Very well).
  The overall range of possible scores is 5 to 25, with a higher score indicating a higher level of empathic self-efficacy.
Job Self-efficacy | Pre-intervention, immediately post-intervention, 3-month post-intervention
  Score of Job Self-Efficacy (JSE) was used to assess participants' changes job self-efficacy.
  Each item is rated on a scale, ranging from 1 (Very much disagree) to 6 (Very much agree). Individual item scores are summed to create a total raw score. Raw scores from the items or subscales are summed to form composite scores, with higher scores indicating greater self-efficacy in job-related tasks.

SECONDARY OUTCOMES:
Adaptive Functioning | Pre-intervention, immediately post-intervention, 3-month post-intervention
  General Adaptive Composite (GAC) score of the Adaptive Behavior Assessment System: Third Edition (ABAS-3) was used to assess participants' changes in adaptive functioning skills.
  Raw Scores: Each item within the domains is rated on a 4-point Likert scale, ranging from 0 (Never) to 3 (Always). The ratings are summed to produce raw scores for each domain, which include (1) Conceptual: communication, functional academics, and self-direction; (2) Social: Includes social skills and leisure; (3) Practical: Includes self-care, home living, community use, health and safety, and work.
  Scaled Scores: Raw scores are converted to scaled scores for each domain. Scaled scores typically range from 1 to 19, with a mean of 10 and a standard deviation of 3.
  Composite Score: The scaled scores from the domains are combined to form the GAC, with a mean of 100 and a standard deviation of 15, with a higher score indicating high social functioning.
Psychosocial Functioning | Pre-intervention, immediately post-intervention, 3-month post-intervention
  Score of the Behavior Assessment System for Children: Third Edition (BASC-3) was used to assess participants' changes in adaptive functioning skills.
  Raw Scores: Each item within the domains is rated on a 4-point Likert scale, ranging from 0 (Never) to 3 (Always). The ratings are summed to produce raw scores for each subscale, which include (1) Anxiety; (2) Depression; (3) Withdrawal; (4) Adaptability; (5) Leadership; (6) Executive Functioning; (7) Resiliency.
  T-scores: Raw scores are converted to T-scores to facilitate interpretation. T-scores have a mean of 50 and a standard deviation of 10, with a higher score indicating greater severity of psychosocial impairment.
Work Readiness | Pre-intervention, immediately post-intervention, 3-month post-intervention
  Scaled score of the Stages of Change-Work Participation Scale (SCWPS) was used to assess participants' changes in work readiness.
  Raw Scores: Each item is rated on a 5-point Likert scale ranging from 1 (Strongly disagree) to 5 (strongly agree), and the scores are summed for items corresponding to each stage of change.
  Stage Classification: The sum of scores within each stage helps classify the individual's current stage of readiness for change in work participation.
Anxiety | Pre-intervention, immediately post-intervention, 3-month post-intervention
  Total score of the General Anxiety Disorder-7 (GAD-7) was used to assess participants' changes in anxiety symptoms.
  Items are rated on a 4-point Likert scale, ranging from 0 (Not at all) to 3 (Nearly everyday). Sum the scores for all 7 items to obtain the total score. Total score ranges from 0 to 21, with a higher score indicating higher anxiety.
Depression | Pre-intervention, immediately post-intervention, 3-month post-intervention
  Total score of the Patient Health Questionnaire-9 (PHQ-9) was used to assess participants' changes in depressive symptoms.
  Items are rated on a 4-point Likert scale, ranging from 0 (Not at all) to 3 (Nearly everyday). Sum the scores for all 9 items to obtain the total score. Total score ranges from 0 to 27, with a higher score indicating higher depression.
Life Satisfaction | Pre-intervention, immediately post-intervention, 3-month post-intervention
  Total score of the Satisfaction With Life Scale (SWLS) was used to participants' changes in life satisfaction.
  Items are rated on a 7-point Likert scale, ranging from 1 (Strongly disagree) to 5 (Strongly agree). Sum the scores for all 5 items to obtain the total score. Total score ranges from 5 to 35, with higher score indicating higher depression.

CONTACTS AND LOCATIONS:
Overall Officials: Connie Sung, PhD, Principal Investigator — Michigan State University
Locations (1):
- Michigan State University, East Lansing, Michigan, United States

IPD SHARING:
Plan to Share IPD: No